CLINICAL TRIAL: NCT07285408
Title: Impact of Body Composition, Sarcopenia, Myosteatosis, and Nutritional Status on Recurrence and Progression in Patients With Non-Muscle-Invasive Bladder Cancer: A Prospective Observational Study
Brief Title: Sarcopenia and NMIBC Prognosis Study
Acronym: SARC-NMIBC
Status: Not yet recruiting | Type: Observational
Sponsor: General Hospital Sveti Duh (Other)
Responsible Party: Principal Investigator, Adelina Hrkac, MD, FEBU, General Hospital Sveti Duh
Other Study IDs: KBSD-2025-03-3556; KBSD-URO--2025 (Registry Identifier: KB Sveti Duh Urology Institutional Research Registry)
Record Dates: First submitted 2025-11-30; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Bladder Cancer Cell Transitional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Altered Body Composition / Nutritional Risk: Participants with one or more body composition or nutritional abnormalities, including sarcopenia (low skeletal muscle index), myosteatosis (low skeletal muscle density), obesity (elevated BMI or waist circumference), or malnutrition (NRS ≥ 3 or low serum albumin). These participants will undergo standard TURBT and prospective follow-up to evaluate recurrence and progression of NMIBC.
- Normal Body Composition / No Nutritional Risk: Participants without sarcopenia, myosteatosis, obesity, or malnutrition according to predefined clinical and radiologic criteria. These individuals will also undergo standard TURBT and prospective NMIBC surveillance to allow comparison of recurrence and progression outcomes with the altered body composition group.

SUMMARY:
The goal of this observational study is to evaluate whether body composition abnormalities (sarcopenia, myosteatosis, and obesity) and nutritional status influence the risk of recurrence and progression in adult patients with non-muscle-invasive bladder cancer (NMIBC). The main questions it aims to answer are:

Do sarcopenia, myosteatosis, obesity, or malnutrition increase the likelihood of NMIBC recurrence and progression?

Can clinical, laboratory, and CT-derived body composition parameters serve as predictive biomarkers that improve individualized risk stratification?

Participants will undergo routine clinical and radiologic assessments, including:

* completion of the SARC-F and NRS nutritional screening questionnaires
* anthropometric measurements (BMI, waist circumference)
* laboratory evaluation including serum albumin and testosterone
* CT-based assessment of skeletal muscle index (SMI) and muscle density (SMD)
* standard TURBT and structured follow-up with cystoscopy, cytology, imaging, and clinical evaluations to document recurrence and progression.

DETAILED DESCRIPTION:
Non-muscle-invasive bladder cancer (NMIBC) accounts for approximately 75% of bladder cancer cases and is characterized by a high rate of recurrence and a variable risk of progression. Existing prognostic models, such as EAU and EORTC calculators, incorporate tumor-specific features but do not consider patient-related factors such as body composition or nutritional status. Emerging evidence suggests that sarcopenia, myosteatosis, obesity, and malnutrition may adversely influence oncologic outcomes through mechanisms involving systemic inflammation, impaired immune response, metabolic dysfunction, and reduced physiological reserve. These host-related factors may therefore represent important, yet under-recognized, prognostic biomarkers in NMIBC.

This prospective observational cohort study aims to determine whether clinical and radiologic measures of body composition and nutritional status are associated with the risk of recurrence and progression in patients with NMIBC. Preoperative assessment will include SARC-F screening for sarcopenia, NRS screening for nutritional risk, anthropometric measurements (BMI and waist circumference), serum albumin and testosterone measurement, and CT-based quantification of skeletal muscle index (SMI) and skeletal muscle density (SMD). Tumor-related variables including stage, grade, presence of carcinoma in situ, variant histology, lymphovascular invasion, and tumor size and multiplicity will be abstracted from pathology and clinical records. All participants will undergo standard transurethral resection of bladder tumor (TURBT), and postoperative management will follow guideline-recommended NMIBC surveillance schedules based on individual EAU/EORTC risk stratification.

During follow-up, patients will undergo regular cystoscopic evaluations, urine cytology, serial SARC-F and NRS assessments, anthropometric measurements, albumin monitoring, and periodic CT imaging to reassess SMI and SMD. Recurrence and progression events will be documented according to standard clinical criteria.

By identifying clinically meaningful host-related predictors of recurrence and progression, this study may improve individualized risk stratification, inform tailored surveillance strategies, and highlight the need for early identification and correction of adverse body composition and nutritional states in patients with NMIBC.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Histologically confirmed non-muscle-invasive bladder cancer (NMIBC) (Ta, T1, or CIS)
* Scheduled for transurethral resection of bladder tumor (TURBT) as part of standard care
* Able to undergo CT imaging required for assessment of skeletal muscle index (SMI) and skeletal muscle density (SMD)
* Completed preoperative clinical evaluation including: SARC-F, NRS, anthropometric measurements (BMI, waist circumference), serum albumin, and routine laboratory tests
* Able and willing to provide written informed consent

Exclusion Criteria:

* Low-risk NMIBC, as defined by clinical guidelines
* Muscle-invasive bladder cancer (≥ T2) at diagnosis
* Expected survival less than 3 months
* Contraindications to CT imaging (e.g., severe renal dysfunction, contrast allergy if contrast required)
* Age under 18 years
* Inability or unwillingness to adhere to scheduled follow-up
* Any condition that, in the investigator's judgment, would interfere with participation or data integrity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with non-muscle-invasive bladder cancer (NMIBC) undergoing transurethral resection of bladder tumor (TURBT) and guideline-based surveillance at a tertiary urology center. The study population includes individuals with and without body composition and nutritional abnormalities (sarcopenia, myosteatosis, obesity, or malnutrition) who meet eligibility criteria and consent to participate.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2027-07-12 (Estimated); Study Completion 2029-07-09 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 36 months
  Time from TURBT to progression to muscle-invasive bladder cancer (≥ T2) or other defined progression endpoints (CIS emergence, variant histology progression).
Recurrence-Free Survival (RFS) | Up to 36 months
  Time from transurethral resection of bladder tumor (TURBT) to the first documented recurrence of non-muscle-invasive bladder cancer, confirmed by cystoscopy, urine cytology, or pathology.

SECONDARY OUTCOMES:
Impact of Preoperative Skeletal Muscle Index (SMI) on Recurrence Free Survival (RFS) | baseline to 36 months
  Recurrence-free survival according to skeletal muscle index (SMI) measured on baseline computed tomography (CT) images at L3 level (cm²/m²).
Impact of Preoperative Skeletal Muscle Density (SMD) on Recurrence Free Survival (RFS) | baseline to 36 months
  Recurrence-free survival according to skeletal muscle density (SMD) measured in Hounsfield units (HU) on baseline computed tomography (CT) images at L3 level
Impact of Preoperative Body Mass Index (BMI) on Recurrence Free Survival (RFS) | baseline to 36 months
  Recurrence-free survival according to body mass index (BMI) measured at the baseline evaluation (kg/m²)
Impact of Preoperative Nutritional Risk Score (NRS 2002) on Recurrence Free Survival (RFS) | baseline to 36 months
  Recurrence-free survival according to Nutritional Risk Score (NRS 2002) assesed at the baseline evaluation (expressed in points using the standardized NRS-2002 questionnaire)
Overall Survival (OS) | Up to 36 months
  Time from TURBT to death from any cause.
Cancer-Specific Survival (CSS) | Up to 36 months
  Time from TURBT to death specifically attributed to bladder cancer.
Impact of Preoperative Skeletal Muscle Index (SMI) on Progression Free Survival (PFS) | baseline to 36 months
  Progression-free survival according to skeletal muscle index (SMI) measured on baseline computed tomography (CT) images at L3 level (cm²/m²).
Impact of Preoperative Skeletal Muscle Density (SMD) on Progression Free Survival (PFS) | baseline to 36 months
  Progression-free survival according to skeletal muscle density (SMD) measured in Hounsfield units (HU) on baseline computed tomography (CT) images at L3 level
Impact of Preoperative Body Mass Index (BMI) on Progression Free Survival (PFS) | baseline to 36 months
  Progression-free survival according to body mass index (BMI) measured at the baseline evaluation (kg/m²)
Impact of Preoperative Nutritional Risk Score (NRS 2002) on Progression Free Survival (PFS) | baseline to 36 months
  Progression-free survival according to Nutritional Risk Score (NRS 2002) assesed at the baseline evaluation (expressed in points using the standardized NRS-2002 questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Adelina Hrkac, MD, Principal Investigator — Klinička bolnica "Sveti Duh", Zavod za urologiju

IPD SHARING:
Plan to Share IPD: No